CLINICAL TRIAL: NCT02299583
Title: Protocol for a Controlled Trial of Early Intervention With Children and Adolescents Exposed to Nonrelational Traumatic Events Comparing Trauma-informed and Usual Health Care Practice
Brief Title: Controlled Trial of Early Intervention With Children and Adolescents Exposed to Nonrelational Traumatic Events
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carolina Magdalene Maier (Other)
Collaborators: The Egmont Foundation (Unknown); Ramboll Group (Unknown)
Responsible Party: Sponsor-Investigator, Carolina Magdalene Maier, cand.scient.soc., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: f-22834-02
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Posttraumatic Stress Disorder; Depression; Anxiety
Keywords: prevention; early intervention; trauma-informed practice
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preventive intervention (Experimental): In this arm HCPs will conduct a trauma-informed early intervention with children and families after exposure to potentially traumatic events (PTE).
  Interventions: Other: Preventive intervention trauma-informed early intervention
- Control group (No Intervention): There will be no intervention in this arm. The outcome will show the efficiency of usual care.

INTERVENTIONS:
Other: Preventive intervention trauma-informed early intervention — Every department appoints 2-4 health care professionals as child welfare officers (CWOs) who will be responsible for carrying out the intervention at the department. Whenever a child or adolescent is present in the department a CWO will be send for. The intervention consists of four distinct elements: 1) A standardized plan of action for the appointed health care CWOs on how to conduct trauma-informed health care for children and their families shortly after exposure to a PTE, 2) a training program for CWOs on trauma-informed support and communication with children and their families, 3) a supervision program for the CWOs, and 4) three psychoeducational booklets for young children, older children, and parents. The booklets will be given to the families by the CWOs.
  Arms: Preventive intervention

SUMMARY:
Background: International studies have shown that a substantial number of children and adolescents are exposed to potentially traumatic events. Many of these children and adolescents, some of whom will experience posttraumatic stress disorder (PTSD), are submitted to health care departments shortly after exposure as the most common types of traumatic events are accidental injury, serious somatic illness or death of someone close. There has been some research on early psychological interventions for prevention and treatment of PTSD. However, very little research has examined the efficacy of trauma-informed practice among health care professionals (HCPs). The present trial aims to evaluate and compare trauma-informed health care with usual practice.

Methods/Design: The primary clinical question under investigation is the efficacy of an early, trauma-informed intervention for the prevention of PTSD in children and adolescents following exposure to a potentially traumatic event. The trail compares a standardized trauma-informed practice with usual care (no intervention) in health care departments receiving children and adolescents after exposure to determine if trauma-informed care is associated with a reduction in psychological outcome measures over time. Specifically, the investigators examine the efficacy of health care professional's active use of trauma-informed standards of action and a trauma training program for HCPs in the intervention group. The primary outcome will be a reduction in trauma, anxiety and depressive symptoms on self-reports in the active intervention compared to usual care.

Discussion: This trial will be the first controlled trial to examine a trauma-informed intervention carried out by HCPs. It will provide the first evidence on the efficacy of health care delivered by trauma-educated HCPs using trauma-informed standards of action. A successful implementation of this protocol will support the thesis that prevention of PTSD among children and adolescents benefits from a focus on the practice of HCPs. If efficacious, the results will be a call for future research to extend the investigation of interventions from psychological treatment to HCP-based care.

DETAILED DESCRIPTION:
Background

A significant number of children and adolescents have been exposed to potentially traumatic events (PTEs). American and Australian studies report a prevalence of about 20-25% of high magnitude traumatic events among adolescents. A Danish study of four Nordic countries found that 90 % of adolescents with a mean age of 14.5 years had been exposed to at least one low magnitude traumatic event.

A potentially traumatic event may be either relational such as sexual or physical abuse or nonrelational such as illness, motor vehicle accident or fire. The incidence of nonrelational trauma is very high in children and adolescents with accidental injuries being the largest cause of morbidity and mortality among children in the United States as well as in Denmark. Although many children and adolescents demonstrate great resilience or appear to be only briefly affected by nonrelational traumatic events a significant minority of young people will develop posttraumatic stress disorder (PTSD), posttraumatic stress symptoms (PTSSs) or other psychological difficulties following exposure to trauma.

Accidental injury is the most common type of trauma. Researchers report prevalence rates of PTSD among children and adolescents in road traffic accidents ranging from 6% to 35%. Rates of PTSSs (also termed subclinical, subthreshold or partial PTSD) range from 11% to 50%6-14. These rates are important since recent research has indicated only minor differences in terms of distress and impairment between children meeting full and partial criteria for PTSD.

The diagnosis of medical illness such as cancer or diabetes has also been shown to cause PTSD in some children and adolescents with prevalence rates of 5.4% for diabetes and of 10% to 18% for cancer. A recent meta-analysis of prevalence related to both injury and illness reported average prevalence rates of PTSD related to injury ranging from 0% to 37.5%, with a mean of 19.82%, and rates in ill youth ranging from 0% to 32%, with a mean of 12.04%.

Preventive interventions for children and adolescents

Given the high prevalence rates of exposure and the likewise high prevalence rates of PTSD and PTSSs after PTEs there is a pressing need for preventive interventions that decrease the risk of PTSD. In a recent systematic review by Forman-Hoffman et al. (2013) of interventions for children exposed to nonrelational traumatic events 6 different interventions based exclusively on exposure were identified. These included trauma-focused cognitive-behavioural therapy child and family traumatic stress intervention (CFTSI), 2 different school interventions with elements of CBT, early psychological intervention and a propranolol study. The two latter studies found no improvement in outcomes, the remaining 4 interventions found some improvement with regards to PTSD, severity of PTSD and PTSSs.

Another recent meta-analysis by Kramer (2011) reviewing early psychological interventions in children and adolescents after single trauma included seven studies (two of which reappeared in the above mentioned review). These included CFTSI, school-based interventions, early psychological interventions, and two interventions based exclusively on psychoeducational information provision. The authors concluded that intervention effects regarding PTSSs and PTSD were small or non-significant but found promising beneficial tendencies with regards to dissociation, anxiety and, to some extent, arousal.

Overall, the empirical literature has not supported the effectiveness of early psychological interventions such as psychological debriefing and single-session psychological intervention on preventing PTSD and PTSSs in children. These results are consistent with a Cochrane review by Rose 2002 of the effects of psychological debriefing for preventing PTSD in adults. However, school-based and family-focused interventions, as well as stepped-procedure and multiple-session psychological interventions have shown promising results.

In conclusion, the current outcomes of the empirical research suggest early interventions that include the following elements31: age-appropriate psychoeducation, the provision of individual coping skills, parental involvement, social support, risk-assessment, multiple sessions and trauma exposure.

The modest results of early psychological interventions suggest a need for a broader perspective on preventive interventions for children and adolescents exposed to nonrelational trauma. Despite the variety of interventions evaluated by the studies included in the two cited reviews none of the studies focused on the practice of health care professionals. This study is the first to conduct a controlled trial of a standardized preventive intervention conducted by health care professionals. The intervention to be evaluated in this study includes all of the above mentioned empirically supported elements except multiple sessions and trauma exposure.

Trauma-informed health care

The concept of trauma-informed practice has been advocated by institutions and researchers in diverse areas such as psychology, mental health care, education, child welfare, first responders, juvenile justice, and health care. The main aim of trauma-informed practice is to create systematic approaches within these areas to develop evidence-based services that address the impact of trauma on the children they serve37. This study will provide evidence on the impact of the practice of HCPs on symptoms, coping and social functioning of children, adolescents and their families who have been exposed to nonrelational trauma. It investigates the effects of educating HCPs in trauma-informed practice and the effects of a standardized trauma-informed plan of action implemented in health care departments working with children and adolescents.

Design of the trial

This study is designed as a controlled trial with one active intervention and one comparison. The study will be conducted across 19 health care departments in 7 hospitals in the Capitol Region of Denmark. There will be two measurement occasions: one assessment 4 weeks after exposure and one follow-up 6 months after exposure. The trial will run over 18 months. During the first 12 months the intervention will run in 12 of the participating departments while the other 8 departments will function as a control group. During the last 6 months the intervention will run in all nineteen departments thus expanding the sample size of the intervention group. Since the intervention is carried out by health care professionals shortly after exposure, the children in the control group will not receive intervention at any point.

Because the intervention investigated in this trial is conducted by HCPs as an integrated part of their general practice (as opposed to a specific treatment program), it was neither practically possible nor ethically sound to design the allocation of participants in the control and intervention group as a randomization of subjects. For this reason, the allocation was done, not on a subject level, but on the level of departments. This precluded an actual randomization of the trial. However, it should be noted that the allocation of the departments is done before the intervention and thus prior to the recruitment of participants. This means that the allocation of subjects was predetermined in advance of their admission to the hospital. This prevents some of the bias associated with the lack of randomization. In the allocation of departments the best possible match of patient groups was pursued.

It is the hypotheses of this study that: The children and adolescents who receive the intervention, compared to participants in the control group, will demonstrate greater reduction in posttraumatic stress, anxiety and depressive symptoms and higher ratings on positive cognitive coping skills and social functioning.

Sample Size and Power Calculation

Given that this is the first trial to examine the effect of a trauma-informed intervention conducted by HCPs as part of their general health care practice, calculations of power were very limited. Furthermore, effect sizes from related trials such as early psychological interventions and interventions based on information provision have been small or non-significant. Given these limitations, however, calculations of power were conducted on the basis of the available evidence.

Results from a study by Kenardy et al. (2008) on an information-provision intervention had an effect size of 0.63 (between groups) on child anxiety. In a similar study by Cox et al. (2010) effect size on child anxiety was 0.33. Based on the results from Cox et al. (2010) a power analysis revealed that 115 families per group (N = 230) will result in 80% power for detecting a significant difference between the intervention and the control group at the 5% significance level. However, with an estimated 25% attrition rate over the assessment time periods, a total of 290 families should be aimed at to be recruited for the study.

Another power analysis was conducted to calculate the power given a specific sample size. This was done because the participating departments are required to include all eligible families presented to the departments during the intervention period. It was estimated that each department would receive two eligible participants per month. Because of the difference in size between the intervention group and the control this resulted in a sample size of 516 for the intervention group and 168 for the control group (N = 684). With an estimated 25 % attrition rate these numbers amount to 387 for the intervention group and 126 for the control group (N = 513). A post hoc power calculation resulted in 94 % power with an effect size of 0.33 and a 5 % significance level.

Statistical Considerations

Prior to statistical analysis of outcomes, the control group and the intervention group will be compared for pre-intervention equivalence on demographic information and type of PTE. If significant differences are identified, this will be taken into account by including these variables as covariates in outcome analyses. The outcome data will be analysed and reported in terms of statistical significance of difference between intervention and control group in change over time on outcome, clinical significance of the change, and effect sizes. The analysis will be performed by researchers who have not been involved in assessing eligibility of participants, collection of data or entering of data.

Primary analysis will be undertaken on an intention-to-treat (ITT) basis, including all participants who have received intervention or have been registered to the control group, regardless of withdrawal from the study. The data will be analysed with a mixed effects model, which is able to include participants whose data may be partly missing. Analysis of covariance will be conducted with three pairs of outcome: 1) child and parent outcome, 2) symptom outcome and coping outcome, and 3) symptom outcome and social functioning outcome. Other outcomes such as demographics and types of PTE will be described.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 8 and 18 years
* Admission to hospital for accidental injury involving danger to life, serious injury or impairment
* Admission to hospital for acute illness involving danger to life, serious injury or impairment
* Sudden severe impairment of medical condition
* Admission of parent or sibling to hospital for accidental injury involving danger to life, serious injury or impairment
* Admission of parent or sibling to hospital for acute illness involving danger to life, serious injury or impairment
* Sudden severe impairment of parental or sibling medical condition
* Consent to participate in the study

Exclusion Criteria:

* Parent's Danish insufficient for questionnaire completion
* Developmental delay or mental retardation in the child
* Moderate to severe head injury or posttraumatic amnesia following the accident
* Injury due to physical or sexual abuse (intentional injury)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 684 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Severity of posttraumatic stress symptoms (Children's Revised Impact of Event Scale.) | 4 weeks after the traumatic event
  The child assessment will be administered with the Children's Revised Impact of Event Scale.
  The parent primary outcome measure will be assessed with the Impact of Event Scale.
Severity of posttraumatic stress symptoms (Children's Revised Impact of Event Scale.) | 6 months after the traumatic event
  The child assessment will be administered with the Children's Revised Impact of Event Scale.
  The parent primary outcome measure will be assessed with the Impact of Event Scale.
Change from baseline in severity of posttraumatic stress symptoms at 6 months (Children's Revised Impact of Event Scale.) | 4 weeks and 6 months after the traumatic event
  The child assessment will be administered with the Children's Revised Impact of Event Scale.
  The parent primary outcome measure will be assessed with the Impact of Event Scale.
Severity of anxiety symptoms (Revised Child Anxiety and Depression Scale.) | 4 weeks after the traumatic event
  The assessment will be administered with the Revised Child Anxiety and Depression Scale.
Severity of anxiety symptoms (Revised Child Anxiety and Depression Scale.) | 6 months after the traumatic event
  The assessment will be administered with the Revised Child Anxiety and Depression Scale.
Change from baseline in severity of anxiety symptoms at 6 months (Revised Child Anxiety and Depression Scale.) | 4 weeks and 6 months after the traumatic event
  The assessment will be administered with the Revised Child Anxiety and Depression Scale.
Severity of depressive symptoms (Revised Child Anxiety and Depression Scale.) | 4 weeks after the traumatic event
  The assessment will be administered with the Revised Child Anxiety and Depression Scale.
Severity of depressive symptoms (Revised Child Anxiety and Depression Scale.) | 6 months after the traumatic event
  The assessment will be administered with the Revised Child Anxiety and Depression Scale.
Change from baseline in severity of depressive symptoms at 6 months (Revised Child Anxiety and Depression Scale.) | 4 weeks and 6 months after the traumatic event
  The assessment will be administered with the Revised Child Anxiety and Depression Scale.

SECONDARY OUTCOMES:
Social functioning of the family (Crisis Support Scale and the WHO-Five Well-being Index.) | 4 weeks after the traumatic event
  The child assessment will be administered with the Crisis Support Scale. The parent secondary outcome measure will be assessed with the Crisis Support Scale and the WHO-Five Well-being Index.
Social functioning of the family (Crisis Support Scale and the WHO-Five Well-being Index.) | 6 months after the traumatic event
  The child assessment will be administered with the Crisis Support Scale. The parent secondary outcome measure will be assessed with the Crisis Support Scale and the WHO-Five Well-being Index.
Change from baseline in social functioning of the family at 6 months (Crisis Support Scale and the WHO-Five Well-being Index.) | 4 weeks and 6 months after the traumatic event
  The child assessment will be administered with the Crisis Support Scale. The parent secondary outcome measure will be assessed with the Crisis Support Scale and the WHO-Five Well-being Index.
Cognitive coping skills of the children and their parents ( Post-traumatic Cognitions Inventory.) | 4 weeks after the traumatic event
  The child assessment will be administered with the Children's Post-traumatic Cognitions Inventory.
  The parent secondary outcome measure will be assessed with the Post-traumatic Cognitions Inventory.
Cognitive coping skills of the children and their parents ( Post-traumatic Cognitions Inventory.) | 6 months after the traumatic event
  The child assessment will be administered with the Children's Post-traumatic Cognitions Inventory.
  The parent secondary outcome measure will be assessed with the Post-traumatic Cognitions Inventory.
Change from baseline in cognitive coping skills of the children and their parents at 6 months ( Post-traumatic Cognitions Inventory.) | 4 weeks and 6 months after the traumatic event
  The child assessment will be administered with the Children's Post-traumatic Cognitions Inventory.
  The parent secondary outcome measure will be assessed with the Post-traumatic Cognitions Inventory.

OTHER OUTCOMES:
The families' satisfaction with the intervention program (Intervention Satisfaction Questionnaire) | 4 weeks after traumatic event
  It will be measured through an author developed Intervention Satisfaction Questionnaire, completed by parents and children.
The families' relational coping skills (Relational Coping Questionnaire ) | 4 weeks after the traumatic event
  It will be measured through an author developed Relational Coping Questionnaire covering questions that are not included in the secondary outcome measures.
The families' relational coping skills (Relational Coping Questionnaire ) | 6 months after the traumatic event
  It will be measured through an author developed Relational Coping Questionnaire covering questions that are not included in the secondary outcome measures.
Change from baseline in the families' relational coping skills at 6 months (Relational Coping Questionnaire ) | 4 weeks and 6 months after the traumatic event
  It will be measured through an author developed Relational Coping Questionnaire covering questions that are not included in the secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Lasse P Michelsen, MA, Principal Investigator — Rigshospitalet, Denmark; Ditte B Eriksen, LPsy, Principal Investigator — Rigshospitalet, Denmark; Carolina M Maier, MSc, Study Director — Rigshospitalet, Denmark
Locations (1):
- Hospitals of the Capitol Region of Denmark, Copenhagen, Denmark

REFERENCES:
- [Background] Costello EJ, Erkanli A, Fairbank JA, Angold A. The prevalence of potentially traumatic events in childhood and adolescence. J Trauma Stress. 2002 Apr;15(2):99-112. doi: 10.1023/A:1014851823163. PMID 12013070
- [Background] Cox CM, Kenardy JA, Hendrikz JK. A randomized controlled trial of a web-based early intervention for children and their parents following unintentional injury. J Pediatr Psychol. 2010 Jul;35(6):581-92. doi: 10.1093/jpepsy/jsp095. Epub 2009 Nov 11. PMID 19906829
- [Background] Elklit A, Petersen T. Exposure to traumatic events among adolescents in four nations. Torture. 2008;18(1):2-11. PMID 19289877
- [Background] Hamilton BE, Hoyert DL, Martin JA, Strobino DM, Guyer B. Annual summary of vital statistics: 2010-2011. Pediatrics. 2013 Mar;131(3):548-58. doi: 10.1542/peds.2012-3769. Epub 2013 Feb 11. PMID 23400611
- [Background] Di Gallo A, Barton J, Parry-Jones WL. Road traffic accidents: early psychological consequences in children and adolescents. Br J Psychiatry. 1997 Apr;170:358-62. doi: 10.1192/bjp.170.4.358. PMID 9246255
- [Background] Mirza KA, Bhadrinath BR, Goodyer IM, Gilmour C. Post-traumatic stress disorder in children and adolescents following road traffic accidents. Br J Psychiatry. 1998 May;172:443-7. doi: 10.1192/bjp.172.5.443. PMID 9747409
- [Background] Stallard P, Velleman R, Baldwin S. Prospective study of post-traumatic stress disorder in children involved in road traffic accidents. BMJ. 1998 Dec 12;317(7173):1619-23. doi: 10.1136/bmj.317.7173.1619. PMID 9848900
- [Background] Stallard P, Velleman R, Baldwin S. Psychological screening of children for post-traumatic stress disorder. J Child Psychol Psychiatry. 1999 Oct;40(7):1075-82. PMID 10576537
- [Background] de Vries AP, Kassam-Adams N, Cnaan A, Sherman-Slate E, Gallagher PR, Winston FK. Looking beyond the physical injury: posttraumatic stress disorder in children and parents after pediatric traffic injury. Pediatrics. 1999 Dec;104(6):1293-9. doi: 10.1542/peds.104.6.1293. PMID 10585980
- [Background] McDermott BM, Cvitanovich A. Posttraumatic stress disorder and emotional problems in children following motor vehicle accidents: an extended case series. Aust N Z J Psychiatry. 2000 Jun;34(3):446-52. doi: 10.1080/j.1440-1614.2000.00753.x. PMID 10881968
- [Background] Keppel-Benson JM, Ollendick TH, Benson MJ. Post-traumatic stress in children following motor vehicle accidents. J Child Psychol Psychiatry. 2002 Feb;43(2):203-12. doi: 10.1111/1469-7610.00013. PMID 11902599
- [Background] Landolt MA, Vollrath M, Timm K, Gnehm HE, Sennhauser FH. Predicting posttraumatic stress symptoms in children after road traffic accidents. J Am Acad Child Adolesc Psychiatry. 2005 Dec;44(12):1276-83. doi: 10.1097/01.chi.0000181045.13960.67. PMID 16292120
- [Background] Kassam-Adams N, Winston FK. Predicting child PTSD: the relationship between acute stress disorder and PTSD in injured children. J Am Acad Child Adolesc Psychiatry. 2004 Apr;43(4):403-11. doi: 10.1097/00004583-200404000-00006. PMID 15187800
- [Background] Carrion VG, Weems CF, Ray R, Reiss AL. Toward an empirical definition of pediatric PTSD: the phenomenology of PTSD symptoms in youth. J Am Acad Child Adolesc Psychiatry. 2002 Feb;41(2):166-73. doi: 10.1097/00004583-200202000-00010. PMID 11837406
- [Background] Scheeringa MS, Zeanah CH, Myers L, Putnam FW. New findings on alternative criteria for PTSD in preschool children. J Am Acad Child Adolesc Psychiatry. 2003 May;42(5):561-70. doi: 10.1097/01.CHI.0000046822.95464.14. PMID 12707560
- [Background] Scheeringa MS, Wright MJ, Hunt JP, Zeanah CH. Factors affecting the diagnosis and prediction of PTSD symptomatology in children and adolescents. Am J Psychiatry. 2006 Apr;163(4):644-51. doi: 10.1176/ajp.2006.163.4.644. PMID 16585439
- [Background] Iselin G, Le Brocque R, Kenardy J, Anderson V, McKinlay L. Which method of posttraumatic stress disorder classification best predicts psychosocial function in children with traumatic brain injury? J Anxiety Disord. 2010 Oct;24(7):774-9. doi: 10.1016/j.janxdis.2010.05.011. Epub 2010 May 25. PMID 20541906
- [Background] Landolt MA, Vollrath M, Ribi K, Gnehm HE, Sennhauser FH. Incidence and associations of parental and child posttraumatic stress symptoms in pediatric patients. J Child Psychol Psychiatry. 2003 Nov;44(8):1199-207. doi: 10.1111/1469-7610.00201. PMID 14626460
- [Background] Forman-Hoffman VL, Zolotor AJ, McKeeman JL, Blanco R, Knauer SR, Lloyd SW, Fraser JG, Viswanathan M. Comparative effectiveness of interventions for children exposed to nonrelational traumatic events. Pediatrics. 2013 Mar;131(3):526-39. doi: 10.1542/peds.2012-3846. Epub 2013 Feb 11. PMID 23400617
- [Background] Goenjian AK, Karayan I, Pynoos RS, Minassian D, Najarian LM, Steinberg AM, Fairbanks LA. Outcome of psychotherapy among early adolescents after trauma. Am J Psychiatry. 1997 Apr;154(4):536-42. doi: 10.1176/ajp.154.4.536. PMID 9090342
- [Background] Goenjian AK, Walling D, Steinberg AM, Karayan I, Najarian LM, Pynoos R. A prospective study of posttraumatic stress and depressive reactions among treated and untreated adolescents 5 years after a catastrophic disaster. Am J Psychiatry. 2005 Dec;162(12):2302-8. doi: 10.1176/appi.ajp.162.12.2302. PMID 16330594
- [Background] Berkowitz SJ, Stover CS, Marans SR. The Child and Family Traumatic Stress Intervention: secondary prevention for youth at risk of developing PTSD. J Child Psychol Psychiatry. 2011 Jun;52(6):676-85. doi: 10.1111/j.1469-7610.2010.02321.x. Epub 2010 Sep 24. PMID 20868370
- [Background] Berger R, Pat-Horenczyk R, Gelkopf M. School-based intervention for prevention and treatment of elementary-students' terror-related distress in Israel: a quasi-randomized controlled trial. J Trauma Stress. 2007 Aug;20(4):541-51. doi: 10.1002/jts.20225. PMID 17721962
- [Background] Berger R, Gelkopf M. School-based intervention for the treatment of tsunami-related distress in children: a quasi-randomized controlled trial. Psychother Psychosom. 2009;78(6):364-71. doi: 10.1159/000235976. Epub 2009 Sep 8. PMID 19738402
- [Background] Gelkopf M, Berger R. A school-based, teacher-mediated prevention program (ERASE-Stress) for reducing terror-related traumatic reactions in Israeli youth: a quasi-randomized controlled trial. J Child Psychol Psychiatry. 2009 Aug;50(8):962-71. doi: 10.1111/j.1469-7610.2008.02021.x. Epub 2008 Dec 22. PMID 19207621
- [Background] Zehnder D, Meuli M, Landolt MA. Effectiveness of a single-session early psychological intervention for children after road traffic accidents: a randomised controlled trial. Child Adolesc Psychiatry Ment Health. 2010 Feb 8;4:7. doi: 10.1186/1753-2000-4-7. PMID 20181120
- [Background] Nugent NR, Christopher NC, Crow JP, Browne L, Ostrowski S, Delahanty DL. The efficacy of early propranolol administration at reducing PTSD symptoms in pediatric injury patients: a pilot study. J Trauma Stress. 2010 Apr;23(2):282-7. doi: 10.1002/jts.20517. PMID 20419738
- [Background] Kramer DN, Landolt MA. Characteristics and efficacy of early psychological interventions in children and adolescents after single trauma: a meta-analysis. Eur J Psychotraumatol. 2011;2. doi: 10.3402/ejpt.v2i0.7858. Epub 2011 Dec 15. PMID 22893820
- [Background] Poijula S, Dyregrov A, Wahlberg KE, Jokelainen J. Reactions to adolescent suicide and crisis intervention in three secondary schools. Int J Emerg Ment Health. 2001 Spring;3(2):97-106. PMID 11508571
- [Background] Stallard P, Velleman R, Salter E, Howse I, Yule W, Taylor G. A randomised controlled trial to determine the effectiveness of an early psychological intervention with children involved in road traffic accidents. J Child Psychol Psychiatry. 2006 Feb;47(2):127-34. doi: 10.1111/j.1469-7610.2005.01459.x. PMID 16423143
- [Background] Kenardy J, Thompson K, Le Brocque R, Olsson K. Information-provision intervention for children and their parents following pediatric accidental injury. Eur Child Adolesc Psychiatry. 2008 Aug;17(5):316-25. doi: 10.1007/s00787-007-0673-5. Epub 2008 Mar 18. PMID 18350366
- [Background] Rose S, Bisson J, Churchill R, Wessely S. Psychological debriefing for preventing post traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2002;(2):CD000560. doi: 10.1002/14651858.CD000560. PMID 12076399
- [Background] Regan K. Trauma informed care on an inpatient pediatric psychiatric unit and the emergence of ethical dilemmas as nurses evolved their practice. Issues Ment Health Nurs. 2010 Mar;31(3):216-22. doi: 10.3109/01612840903315841. PMID 20144033
- [Background] Azeem MW, Aujla A, Rammerth M, Binsfeld G, Jones RB. Effectiveness of six core strategies based on trauma informed care in reducing seclusions and restraints at a child and adolescent psychiatric hospital. J Child Adolesc Psychiatr Nurs. 2011 Feb;24(1):11-5. doi: 10.1111/j.1744-6171.2010.00262.x. PMID 21272110
- [Background] Layne CM, Strand V, Popescu M, Kaplow JB, Abramovitz R, Stuber M, Amaya-Jackson L, Ross L, Pynoos RS. Using the core curriculum on childhood trauma to strengthen clinical knowledge in evidence-based practitioners. J Clin Child Adolesc Psychol. 2014;43(2):286-300. doi: 10.1080/15374416.2013.865192. Epub 2014 Jan 31. PMID 24484506
- [Background] Mallon GP. Trauma informed child welfare practice--remembering Robert. Child Welfare. 2011;90(6):7-10. No abstract available. PMID 22533038
- [Background] Ursano RJ, Benedek DM, Engel CC. Trauma-informed care for primary care: the lessons of war. Ann Intern Med. 2012 Dec 18;157(12):905-6. doi: 10.7326/0003-4819-157-11-201212040-00542. No abstract available. PMID 22964876
- [Background] Jeggesen A, Gudmundsdóttir DB, Elklit A: Posttraumatic stress disorder in adolescent and Young adult survivors of childhood cancer. Nordic Psychology 2012, 64;4:291-302.
- [Background] Kahana SY, Feeny NC, Youngstrom EA, Drotar D: Posttraumatic Stress in Youth Experiencing Illnesses and Injuries: An Exploratory Meta-Analysis. Traumatology 2006; 12; 148-161
- [Background] Ko SJ, Ford JD, Kassam-Adams N, Berkowitz SJ, Wilson C, Wong M: Creating Trauma-Informed Systems: Child Welfare, Education, First Responders, Health Care, Juvenile Justice. Professional Psychology: Research and Practice 2008, 39;4:396-404
- [Background] Steel W, Malchiodi, CA: Trauma-Informed Practices With Children and Adolescents. Routledge, New York 2012
- [Background] Conners-Burrow NA, Kramer TL, Sigel BA, Helpenstill K, Sievers C, McKelvey L: Trauma-informed care training in a child welfare system: Moving it to the front line. Children and Youth Services Review 2013, 35;11:1830-1835
- [Background] Kramer TL, Sigel BA, Conners-Burrow NA, Savary PE, Tempel A: A statewide introduction of trauma-informed care in a child welfare system. Children and Youth Services Review 2013, 35:19-24
- [Background] Ford, JD, Blaustein, ME: Systemic Self-Regulation: A Framework for Trauma-Informed Services in Residential Juvenile Justice Programs. Journal of Family Violence 2013, 28;7:665-677